CLINICAL TRIAL: NCT00828906
Title: DuoTrav® Eye Drops As Replacement Therapy Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DART-2
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-07

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; IOP; DuoTrav
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Duotrav

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): DuoTrav
  Interventions: Drug: DuoTrav

INTERVENTIONS:
Drug: DuoTrav — DuoTrav Eye Drops

SUMMARY:
To evaluate the effectiveness of DuoTrav Eye Drops in gaining or maintaining control of target Intraocular Pressures (tIOP) in patients diagnosed with, and being treated for, open-angle glaucoma (OAG) or ocular hypertension (OH).

ELIGIBILITY:
Inclusion Criteria:

* Patients with OAG or OH for whom single agent therapy provides insufficient intraocular pressure reduction

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Intra Ocular Pressure | visit 1, Visits 2-3, Visits 6-8

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon for Trial Locations, Beijing, China